CLINICAL TRIAL: NCT03775642
Title: Debunking Myths About Contraceptive Safety Among Women in Kingston, Jamaica
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: FHI 360 (Other); Epidemiology Research and Training Unit of the Jamaica Ministry of Health (Unknown); The University of The West Indies (Other)
Responsible Party: Principal Investigator, Maria F. Gallo, PhD, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017B0412
Record Dates: First submitted 2018-12-11; First posted 2018-12-14 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Contraception Behavior
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention video (Experimental): The intervention video will employ debiasing strategies to correct women's misinformation about the safety of the IUD and implant safety.
  Interventions: Behavioral: Intervention video
- Control video (Placebo Comparator): The video for the control arm will consist of an existing, public-use video on a non-contraception topic of similar duration.
  Interventions: Behavioral: Control video

INTERVENTIONS:
Behavioral: Intervention video — The intervention video will employ the debiasing strategies. It will avoid directly articulating contraception-related myths, but instead will provide a limited number of alternative explanations related to IUD and implant safety.
  Arms: Intervention video
Behavioral: Control video — The video for the control arm will consist of an existing, public-use video on a non-contraception topic of similar duration
  Arms: Control video

SUMMARY:
The primary hypothesis is that the intervention video - based on strategies from cognitive psychology - can correct women's misinformation about long-acting reversible contraception (LARC) and result in higher use of LARC. While there are no direct benefits to participants from being in the study, the research could benefit women in general by providing evidence to help prevent unintended pregnancy. Unlike many interventions that are not feasible for scaling up once shown to be effective in changing people's behavior, the proposed intervention has been carefully designed to impose a low burden to clinic staff and require few resources for translating to wider use. Thus, the investigators expect the intervention to have high potential for influencing clinical care and research for addressing the overall goal of reducing unintended pregnancy.

DETAILED DESCRIPTION:
The investigators will conduct a randomized trial (RT) of consenting adult women (N=220) to test the effectiveness of the final intervention video.

Participants in the RT will complete the "Enrollment Questionnaire" and then will be randomized to either watch a short video on 1) debiasing about LARC safety (intervention arm; n=110) or 2) vector control (control arm; n=110) (Figure 2). Participants then will have the option of receiving routine contraceptive services that follow standard care. After three months, trained interviewers will contact participants to administer the short "Follow-up Questionnaire" via telephone. To corroborate participant reporting of contraception use during follow-up, the investigators also will extract data on LARC use from participant medical records.

ELIGIBILITY:
Inclusion Criteria:

* present at the Comprehensive Health Centre;
* 18-25 years of age; and
* sexually active (defined as ≥1 penile-vaginal act in past month);

Exclusion Criteria:

* known to be pregnant;
* sterilized;
* breastfeeding;
* currently using the IUD or implant; or
* want pregnancy in the next 12 months

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 225 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
Self-reported initiation of LARC (dichotomous variable for either IUD or implant use vs. neither use) | within 3 months of enrollment
  Based on survey question on use of the IUD (y/n) and implant (y/n)

SECONDARY OUTCOMES:
Self-reported belief about IUD safety | 3 months after enrollment
  "Do you think the IUD is very safe, mostly safe, mostly unsafe, or very unsafe?" Responses will be coded as 1-4 (in the order presented) and used in a regression model to determine whether the values differ by randomization arm.
Self-reported belief about implant safety | 3 months after enrollment
  "Do you think the implant is very safe, mostly safe, mostly unsafe, or very unsafe?" Responses will be coded as 1-4 (in the order presented) and used in a regression model to determine whether the values differ by randomization arm.
Self-reported attitudes toward LARC-related bleeding patterns | 3 months after enrollment
  "How do you feel about your bleeding pattern?" Response options consist of "very satisfied, satisfied, neutral, unsatisfied, very unsatisfied." Responses will be coded as 1-5 (in the order presented) and used in a regression model to determine whether the values differ by randomization arm

CONTACTS AND LOCATIONS:
Overall Officials: Maria F Gallo, PhD, Principal Investigator — Ohio State University
Locations (1):
- Epidemiology Training Unit, Kingston, Jamaica

IPD SHARING:
Plan to Share IPD: Undecided